CLINICAL TRIAL: NCT05774990
Title: Incidence and Risk Factors for Invasive Mold Infections in Children During First-Line Chemotherapy for Primary Acute Leukemia: Protocol for a National Retrospective Cohort Study
Brief Title: Study Protocol: Study on Incidence and Risk Factors of Mold Infections in Children During Leukemia Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Odense Patient Data Explorative Network (Other)
Responsible Party: Sponsor
Other Study IDs: 22/15850
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Leukemia, Myeloid, Acute; Acute Lymphoblastic Leukemia
Keywords: leukemia; childhood; myeloid; lymphoblastic; pediatric; invasive; mold; aspergillus
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to evaluate the occurrence, mortality, and risk factors for invasive mold infections (IMI) in children treated with chemotherapy for acute leukemia in Denmark. The study will be a retrospective nationwide survey study of all children who received first-line chemotherapy for acute leukemia from 2008 to 2022 in Danish pediatric oncology units. The study population will include approximately 800 children under the age of 18. Data will be collected from medical records, hospital databases, and national databases. When the IMI subgroup has been identified, this will be compared to the leukemic group that did not develop IMI. Statistical analysis can then determine the occurrence, mortality rate, and possible IMI risk factors.

DETAILED DESCRIPTION:
Chemotherapy can weaken children's immune system, making them vulnerable to infections, including invasive mold infections (IMI), caused mainly by Aspergillus spp. The at-risk population for IMI in children with acquired immunodeficiency is patients with prolonged granulocytopenia due to hematologic malignancies treated with chemotherapy or allogeneic hematopoietic stem cell transplantation (HSCT) recipients and children receiving long-term corticosteroid treatment. Incidences and mortality rates are often reported as high.

In a retrospective cohort study, we aim to obtain an epidemiological overview of IMI in children receiving first-line treatment for acute myelogenous leukemia (AML) and acute lymphoblastic leukemia (ALL) in Denmark from 2008 to 2022 and identify possible risk factors, including treatment-related adverse effects.

Objectives

1. To determine and compare the incidence of IMI in childhood AML and ALL during first-line chemotherapy in Denmark.
2. To determine and compare the mortality of IMI in childhood AML and ALL during first-line chemotherapy in Denmark.
3. To explore risk factors for IMI in childhood AML and ALL during first-line chemotherapy in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years at the time of inclusion
* Received first-line treatment for ALL or AML
* Treatment at a Danish tertiary pediatric oncology unit (Rigshospitalet, Aarhus University Hospital, Odense University Hospital, and Aalborg University Hospital)
* Treatment initiation January 1st, 2008, to December 31st, 2022

Exclusion Criteria:

* Not meeting inclusion criteria

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any patient (<18 years) who initiated first-line chemotherapy against primary ALL or AML at any of the four Danish pediatric oncology departments from January 1st, 2008, to December 31st, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of invasive mold infection in childhood AML and ALL in Denmark | Up to three years
  The number of subjects in the cohort infected with an invasive mold during leukemia treatment period as defined by the European Organization for Research and Treatment of Cancer Mycoses study group (EORTC/MSG) criteria
Mortality form invasive mold infection in childhood AML and ALL in Denmark. | Up to three years
  The number of subjects in the cohort dying from an invasive mold infection during their leukemia treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Møller Duus, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Rasmus Møller Duus, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie the results in a future publication will be made publicly available in an anonymized form.
Supporting Information: Study Protocol
Time Frame: The study protocol will be available before collecting participant data. The anonymized participant data will be made available as supplementary material simultaneously with the publication of the article.
Access Criteria: All who have access to the article can access the participant data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT05774990/Prot_SAP_001.pdf